CLINICAL TRIAL: NCT01275573
Title: High Frequency rTMS (Repetitive Transcranial Magnetic Stimulation) Effect Applied on Primary Cortical Motor, on Nociceptive Perception Thresholds in Parkinson's Disease Patients: a Physiopathology Study
Brief Title: Evaluation of the Effect of Repetitive Transcranial Magnetic Stimulation in Pain Perception in Parkinson's Disease
Acronym: rTMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 09 155 02
Record Dates: First submitted 2010-12-10; First posted 2011-01-12 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson's Disease
Keywords: Repetitive Transcranial Magnetic Stimulation; pain threshold; Parkinson's disease; Pain threshold in Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- healthy volunteers (Other): All the patients and healthy volunteers will receive high frequency Repetitive Transcranial Magnetic Stimulation and placebo stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- painful Parkinson's disease patients (Other): All the patients and healthy volunteers will receive high frequency Repetitive Transcranial Magnetic Stimulation and placebo stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- painless Parkinson's disease patients (Other): All the patients and healthy volunteers will receive high frequency Repetitive Transcranial Magnetic Stimulation and placebo stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation will be applied on the contralateral primary cortical motor on the painful side for the Parkinson's disease patients and on the left primary cortical motor for the healthy volunteer. The stimulation frequency will be 20 Hz during 26 min with an intensity stimulation equal of 95% of the motor threshold.
  Other Names: non applicable

SUMMARY:
Pain is a frequent symptom in Parkinson's disease. Previous studies have shown that pain perception was altered in Parkinson's disease patients and could be related to nociceptive cortical area hyperactivation. Repetitive Transcranial Magnetic Stimulation is an electrophysiological tool which can modify cortical excitability. Its efficacy was demonstrated in neuropathic pain. This is a randomized, double blind cross-over study. In this study, subjective pain threshold (using thermal stimulation (Thermotest)).will be evaluated in 3 groups of subjects: healthy volunteers, painful Parkinson's patients and pain free Parkinson's disease patients. Each group will receive a high frequency Repetitive Transcranial Magnetic Stimulation and placebo stimulation in different order with a gap of one week.

The investigators supposed that a 20 Hz Repetitive Transcranial Magnetic Stimulation session with an infraliminary intensity on the primary cortical motor, modulating nociceptive cortical areas activity, could modify the nociceptive threshold perception in Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patients with clinical diagnosis of Parkinson's disease according to the criteria of the UKPDSBB
* Parkinson's disease patients with a score≤3 on the Hoehn and Year scale
* Patients treated with dopaminergic antiparkinsonian drugs (L-DOPA, dopamine agonists,ICOMT…)
* Patients with or without neuropathic pain induced by Parkinson's disease
* Patients without personal or familial epilepsy episode history
* Patients from 50 to 80 years old (male or female)
* Patients affiliated to a social protection program
* Patient with an informed consent given

For Healthy volunteers

* Subjects from 50 to 80 years old (male or female)
* Subjects without any serious evolutionary pathology or any clinical significant treatment
* Subjects without chronic pain or disease which can induce neuropathic pain
* Subjects without personal or familial epilepsy episode history
* Subjects affiliated to a social protection program
* Subjects with an informed consent given

Exclusion Criteria:

For patients:

* Patients suffering from an other pathology causing chronic pain (rheumatic disease, traumatic or orthopaedic pathologies…)
* Parkinson's disease patients with a score>3 on the Hoehn and Yahr scale
* Patients with important tremors during a OFF conditions
* Patients suffering from a cancer
* Patients with a neuroleptic treatment
* Patients under tutelage, curatella or law protection
* Patients included in an other clinical study
* Patients unable to fulfil scales of the study
* Patients with personal or familial epilepsy episode history
* Contraindication of IRM
* Pregnant women

For Healthy volunteers:

* Subjects with serious evolutionary pathology or any clinical significant treatment
* Subjects with chronic pain or disease which can induce neuropathic pain
* Subjects with personal or familial epilepsy episode history
* Contraindication of IRM
* Pregnant women
* Subjects under tutelage, curatella or law protection
* Subjects included in an other clinical study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change of subjective pain threshold determined using thermal stimulation (Thermotest) with the method of levels after rTMS session | D1 T0, D1 T1h30mn, D7 T0, D7 T1h30mn
  Change from baseline after each Repetitive Transcranial Magnetic Stimulation session (active and placebo)

SECONDARY OUTCOMES:
Analgesic effect of Repetitive Transcranial Magnetic Stimulation using Visual Analogue Scale | D1 T0, D1 T1h30mn, D7 T0, D7 T1h30mn
  Change from baseline after each Repetitive Transcranial Magnetic Stimulation session (active and placebo)
- Clinical evaluation of the severity of the motor handicap of patients using Unified's Parkinson's Disease Rating Scale (UPDRSIII) | D1 T0, D1 T1h30mn, D7 T0, D7 T1h30mn
  Change from baseline after each Repetitive Transcranial Magnetic Stimulation session (active and placebo)
Mood assessment using Visual Analogue Scale | D1 T0, D1 T1h30mn, D7 T0, D7 T1h30mn
  Change from baseline after each Repetitive Transcranial Magnetic Stimulation session (active and placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brefel-Courbon, MD, Principal Investigator — Toulouse Hospital
Locations (1):
- Purpan Hospital, Toulouse, France